CLINICAL TRIAL: NCT02241824
Title: Chronic Opioid Use in Low Back Pain and Lumbar Orthosis Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Geoffrey C. Garth (Other)
Collaborators: VA Long Beach Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Geoffrey C. Garth, Investigator, Aspen Medical Products
Organization: Aspen Medical Products (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIRB# 1273
Record Dates: First submitted 2014-05-26; First posted 2014-09-16 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Lower Back Pain; Chronic Opioid Use
Keywords: Lumbar Orthosis; Lumbar brace

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Elastic abdominal binder (Active Comparator): To evaluate the opioid consumption in chronic low back pain patients on a stable opioid regimen after an intervention of an elastic abdominal binder.
  Interventions: Device: Elastic abdominal binder
- No brace (No Intervention): To evaluate the opioid consumption in chronic low back pain patients on a stable opioid regimen with no brace (control).
- In-elastic lumbar brace (Experimental): To evaluate the opioid consumption in chronic low back pain patients on a stable opioid regimen after an intervention of an in-elastic lumbar brace.
  Interventions: Device: In-elastic lumbar brace

INTERVENTIONS:
Device: In-elastic lumbar brace
  Arms: In-elastic lumbar brace
Device: Elastic abdominal binder
  Arms: Elastic abdominal binder

SUMMARY:
Rationale

* Statement of the Problem. Low back pain is a significant societal problem in the United States, affecting approximately one-fourth of all Americans at any given time. Non-pharmacological therapies have not been well studied although preliminary evidence shows the utilization of bracing may be beneficial in reducing pain and medication usage.
* Hypotheses or Key Question. The investigators hypothesize that the use of an inelastic lumbar brace may decrease opioid use in chronic low back pain patients on a stable opioid regimen. The investigators propose to conduct a randomized controlled study to test our hypothesis.
* Specific Objectives.

AIM 1: To evaluate the opioid consumption in chronic low back pain patients on a stable opioid regimen in a three armed trial, after an intervention of an in-elastic lumbar brace, elastic abdominal binder (standard care), and no brace (control).

AIM 2: To evaluate changes in secondary endpoints such as pain intensity, quality of life, and functional capacity.

Long Term aims: To decrease patient's chronic pain level, improve overall daily function, decrease overall opioid intake and improve quality of life.

DETAILED DESCRIPTION:
Background and Significance

Low back pain (LBP) is a common problem in our society with potential for significant morbidity and mortality. One of the treatments for LBP, opioid therapy, has been increasingly utilized for noncancerous pain,1 and has a 4.2% prevalence in the United States alone.2 The long term use of opioids carries its own risk for adverse events and risk of addiction.3 Thus, with the lack of evidence based research for treatments of LBP, the rising epidemiology of LBP in the US, the rise in cost of medical care, along with the potential risks of opioid therapy, our attention needs to be drawn to find more affordable alternatives.

Our study proposes to evaluate whether an inelastic lumbar brace will reduce chronic opioid use in the chronic low back pain population. The specific aims of this project are to perform a pilot study to assess the feasibility of this project and plan for a larger randomized controlled trial. Additional long-term goals of this study are to assess the effect of an inelastic lumbar brace in a chronic LBP population, and if there is a significant decrease in opioid use and subsequent control or reduction of pain. Secondary endpoints will note improvement in functional outcomes and other quality of life measures. The findings of this preliminary study conducted at the VA facility will provide data to perform a large multi-center randomized controlled trial and prepare for a NIH proposal to study other benefits of inelastic lumbar bracing.

(3) Work Accomplished

(a) New submissions: Preliminary studies have not been conducted yet. (b) Submissions Following Pilot Studies: Sponsored new study

(4) Work Proposed This trial will be a prospective randomized three armed trial of an in-elastic lumbar brace group (BG), elastic abdominal binder (EG), and a control group [no brace] (CG) in the treatment of chronic low back pain patients are prescribed chronic opioid medications with follow-up monitoring up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must satisfy diagnostic criteria for lumbar back pain
* Evidence of lumbar back pain base upon one or more of the following:

  * Lumbar back pain episodes lasting greater than 3 months
  * Has received treatment for recurring nonspecific low back pain
  * Treatment with 3-6 months of stable opioid use.
* Men or women age greater than or equal to 20 years
* Fluency in English

Exclusion Criteria:

* Treatment risk factors including one or more of the following:

  * Unstable or symptomatic cardiac complaints
  * Unstable or symptomatic respiratory complaints
  * Unable to reliably comprehend the protocol or reliably record data
* Pregnancy. A serum pregnancy test must be performed and negative in all women of child bearing potential within 2 weeks prior to enrollment.
* Any medical or psychosocial condition that, in the opinion of the investigator, could jeopardize the subject's participation, and compliance with the study criteria.
* No significant alcohol use (7 or fewer drinks per week).

Ages: 20 Years to 72 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Brace fitting and assessment | Initial visit (month 1 of 12)
  Visit 1: Screening & randomization Study parameters and informed consent will be explained and given to potential participants. If interested, study staff will confirm eligibility and randomize the patient into a group. Patient demographics, medical history and surgical history will be obtained as well as basic vitals. A study team member will then perform the physical function exam, administer the pain assessment, and record current opioid use. Patients will then be fitted for a brace (for those with a brace) and instructed to wear the brace all day, every day except when sleeping or showering. Patients will then be given the packet of quality of life questionnaires and ODI surveys and given ample time to fill them out. Before leaving, patients will schedule the next two phone call checkups and the 3 month visit.
Pain and opioid reduction | Visit 2: (month 3 of 12)
  Visit 2 (3 month visit) When the patient arrives for their appointment, they will leave all bracing in the car so that the physician is blinded when recording information. A study team member will take vitals, review any changes in medication or adverse events and then perform a physical exam documenting range of motion, degree of tender points, and hamstring tightness. The study team member will also record the patients brace wearing compliance, pain assessment and perform a pill count for opioid consumption. The patient will then be asked to fill out the ODI and other quality of life surveys (SF-12 and MPI). Prior to leaving the patient will schedule monthly telephone contacts for the next 8 months as well as their last physical visit at the 12 month time point.
Pain and opioid reduction | Visit 3 (month 12 of 12)
  Visit 3 (12 month visit) When the patient arrives for their appointment, they will leave all bracing in the car so that the physician is blinded when recording information. A study team member will take vitals, review any changes in medication or adverse events and then perform a physical exam documenting range of motion (active and passive), degree of tender points, and hamstring tightness. The study team member will also record the patients brace wearing compliance, pain assessment and perform a pill count for opioid consumption. The patient will then be asked to fill out the ODI and other quality of life surveys (SF-12 and MPI). All patients will be notified that they can keep their brace, if they were given one for the study and that they have completed the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Long Beach VA, Long Beach, California, United States